CLINICAL TRIAL: NCT02653105
Title: Evaluation of the Circulating Concentration of Olfactomédine 4 (OLFM4) in Women With a BRCA1 or 2 Gene Mutation or at High Risk of Developing Breast Cancer, According to the Imaging
Brief Title: Women at Risk of Breast Cancer and OLFM4
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ICO-A-2014-05; 2014-A00305-42 (Other: French Institutional Ethical Committee)
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome
Keywords: High risk of cancer, BRCA1 or 2 mutation, Olfactomedine 4
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OLFM4 (Experimental): Patient have a blood test every 6 months at the same time of the clinical exam planned in the following. The OLFM4 will be dose in the blood sample and the rate of OLFM4 compared to the result of imaging.
  Interventions: Biological: OLFM4

INTERVENTIONS:
Biological: OLFM4 — patient have an additional blood test every 6 months for dosing OLFM4

SUMMARY:
Does the olfactomédine provide an help to limit the number of false positives in the overall imaging balance and limit the number of unnecessary biopsies?

DETAILED DESCRIPTION:
About 5% of breast cancers are associated with the presence of a constitutional genetic alteration. Two genes are being studied: BRCA1 and BRCA2.

The national program for breast cancer screening target women 50 to 74 years but does not include women with significant risk factors. However in identifiable risk situations, breast cancer incidence is increased: and it affects 1 in 4 women with certain risk histological lesions and more than 1 in 2 women carrying a mutation in the BRCA1 or BRCA2 gene.

Studies have shown that the olfactomédine 4 (OLFM4) is highly overexpressed in tumors compared to healthy tissue. The OLFM4 might therefore be a marker for early detection of breast cancer. We wish to determine the positive predictive value of OLFM4 seric dosing of patients at risk with respect to imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* High risk women of breast cancer occurrence defined by the following criteria:

  * Women carrying a genetic mutation BRCA1 or 2 or TP53, entering or already in screening breast IRM
  * Women with a high probability of hereditary predisposition to breast cancer (20% risk at 70 years of breast cancer by BOADICEA model), assessed by the onco-geneticists
* Information of the person and signing the informed consent

Exclusion Criteria:

* Women with a history of breast cancer or in situ
* Person who is not affiliated to a social security scheme or beneficiary of such a regime

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Predictive value of circulating OLFM4 in BRCA1/2 mutation carriers or high-risk women with positive breast imaging | Every 6 months, up to 10 years (120 months)
  The primary objective is to determine the positive predictive value of serum OLFM4 levels in women who are BRCA1 or BRCA2 mutation carriers, or considered at high risk for breast cancer, and who present with a positive imaging workup (including MRI, mammography, and ultrasound) leading to biopsy. The study aims to assess whether OLFM4 can help reduce false positives from imaging and thereby limit unnecessary biopsies. Blood samples will be collected every 6 months over a 10-year period.

CONTACTS AND LOCATIONS:
Overall Officials: Paule AUGEREAU, MD, Principal Investigator — Institut de Cancérologie de l'Ouest - ANGERS
Locations (4):
- France (4):
  - Institut de Cancerologie de l'Ouest, Angers
  - CHU Morvan, Brest
  - Instit de Cancérologie de l'Ouest, Nantes
  - CHBA Hopital Chubert, Vannes

IPD SHARING:
Plan to Share IPD: No